CLINICAL TRIAL: NCT03380247
Title: Multimodal Oral Analgesia for Trauma in the Emergency Department: a Prospective Observational Study of a Nurse-directed Protocol
Brief Title: Multimodal Oral Analgesia for Trauma in the Emergency Department
Acronym: START
Status: Completed | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Collaborators: Mundipharma Pte Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: 38RC17.157; RCB-2017-A01706-47 (Other: Ethic committee [CPP])
Record Dates: First submitted 2017-11-28; First posted 2017-12-21 (Actual); Last update posted 2018-08-03 (Actual); Status verified 2018-08

CONDITIONS: Pain
Keywords: Emergency, trauma pain, analgesia, Methoxyfurane
MeSH Terms: conditions — Pain; Emergencies; Agnosia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The prevalence of pain in the emergency department is estimated between 60% and 78%. However, many studies reported oligo analgesia in about half of patient admitted to the emergency department. The delay before effective analgesia is one of the main causes of oligoanalgesia. The use of nurse-directed protocol allows the administration of analgesic upon admission to the emergency department. Nevertheless the need of intravenous access may delay analgesia. The use of oral form analgesics even with immediate release does not allow effective analgesia before 20 min. Pain management protocol in the emergency reception desk of CHU Grenoble Alpes (CHUGA) includes paracetamol that can be combined with oxycodone tablets depending on the pain intensity. For any mono traumatized it is possible to associate self-administer methoxyflurane inhaler. The pain management protocol is already used in the emergency reception desk of CHU Grenoble Alpes.The different analgesics( paracetamol,oral oxycodone, methoxyflurane) are already administered as part of routine care.The use of these different analgesics means would allow a rapid and adapted effectiveness to the pain intensity. However, there are no data on the efficacy and acceptability of such an early multimodal analgesia protocol in the emergency department.

DETAILED DESCRIPTION:
200 Patients will be included from 8:00 am to 8:00 pm and will receive a multimodal analgesia under the nurse-directed pain management protocol (paracetamol +/- oral oxycodone +/- methoxyflurane) as part of routine medical care.

The pain will be evaluated (Numerical rating scale) prior to the administration and reassessed by a nurse every 5 minutes for 30 minutes and then at 45min and 1 hour after administration of the pain protocol. Satisfaction of patients and caregivers will also be assessed at the end of care.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients : ≥ 18 year and older
* Trauma pain
* NRS≥ 4
* Non- opposition to participate in the study

Exclusion Criteria:

* Trauma with at least one of the following severity criteria:

  * Suspected (from mechanism) or confirmed multiple trauma
  * State of shock
  * Suspected or proven trauma to the thorax (excluding isolated rib fractures with Spo2 ≥ 98%)
  * Suspected or proven Abdominal trauma
  * Suspected or proven pelvic trauma
  * Severe traumatic brain injury
* Altered level of consciousness (Glasgow score < 15)
* Patients who took any analgesic within 4 hours prior to admission (except paracetamol)
* Use of nitrous oxide in the hour before admission
* Patient requiring an intravenous access at admission (e.g. : open fracture displaced)
* Hypersensitivity to one of the molecules of the analgesia protocol
* Known pregnant or likely to be pregnant women at the time of inclusion
* Subject in an exclusion period from another study
* Subjects under tutelage or subjects deprived of liberty
* Patients to be unable to understand the purpose of study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient admitted at the emergency for non-multiple trauma pain
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2017-10-12 (Actual); Primary Completion 2018-07-06 (Actual); Study Completion 2018-07-06 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with a score of less than or equal to 3 on a pain Numeric Rating scale (NRS) (0-10) 15 minutes after inclusion | 15 minutes after inclusion
  NRS scale (0-10)

SECONDARY OUTCOMES:
Secondary efficacy criteria | 15, 30 and 45 min (after inclusion)
  Delay of pain relief defined by a 2 point reduction in the NRS scale (0-10)
Number of patient with 30% reduction in pain intensity | 15,30 and 45 min (after inclusion)
  NRS scale (0-10)
Satisfaction of caregiver and patient | 1h after inclusion
  Patient and caregiver satisfaction evaluated by a visual analog scale (VAS), covering the whole range of analgesic management and in particular each component of multimodal analgesia. The VAS scale ranges are : (not at all satisfied I will not take again - quite satisfied i will take again) for the patient and (not at all satisfied i will not give again - quite satisfied i will give again) for the caregiver

CONTACTS AND LOCATIONS:
Overall Officials: Maxime MAIGNAN, MD PhD, Principal Investigator — University Hospital, Grenoble
Locations (1):
- Emergency Department of University Hospital Grenoble, Grenoble, Auvergne Rhonalpes, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Viglino D, Termoz Masson N, Verdetti A, Champel F, Falcon C, Mouthon A, Mabiala Makele P, Collomb Muret R, Maindet Dominici C, Maignan M. Multimodal oral analgesia for non-severe trauma patients: evaluation of a triage-nurse directed protocol combining methoxyflurane, paracetamol and oxycodone. Intern Emerg Med. 2019 Oct;14(7):1139-1145. doi: 10.1007/s11739-019-02147-8. Epub 2019 Jul 9. PMID 31290084